CLINICAL TRIAL: NCT05655286
Title: The Effectiveness of Silver Diamine Fluoride Treatment With Different Post-treatment Protocols in Arresting Dental Caries in Primary Teeth of Preschool Children
Brief Title: Effectiveness of SDF With Different Post-treatment Protocols in Arresting Dental Caries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chun Hung Chu, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HKU20221001
Record Dates: First submitted 2022-11-30; First posted 2022-12-19 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Dental Caries
Keywords: dental caries; preschool children; silver diamine fluoride
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A- immediately rinse mouth (Experimental): Children are instructed to rinse their teeth with a cup of water containing about 50 ml immediately after SDF treatment. Afterwards, no post-treatment protocol is given to children.
  Interventions: Drug: 38% SDF treatment; Behavioral: rinse mouth immediately after SDF treatment
- Group B- not to rinse for at least 30 minutes (Experimental): Children are instructed not to eat and drink for at least 30 minutes.
  Interventions: Drug: 38% SDF treatment; Behavioral: not to rinse for at least 30 minutes after SDF treatment

INTERVENTIONS:
Drug: 38% SDF treatment — Children with active caries will receive 38% silver diamine fluoride treatment
Behavioral: not to rinse for at least 30 minutes after SDF treatment — After receiving 38% silver diamine fluoride treatment, Children will be asked not to rinse their mouths for at least 30 minutes.
  Arms: Group B- not to rinse for at least 30 minutes
Behavioral: rinse mouth immediately after SDF treatment — After receiving 38% silver diamine fluoride treatment, Children will be asked to rinse their mouths immediately.
  Arms: Group A- immediately rinse mouth

SUMMARY:
To compare the effectiveness of the semi-annual application of 38% SDF with two post-treatment protocols in arresting dental caries in preschool children

DETAILED DESCRIPTION:
Methods: The randomized clinical trial will recruit 254 healthy kindergarten children aged 3-4 years old with caries and with parental consent. All the tooth surfaces with carious lesions will receive the semi-annual application of 38% SDF solution. After the treatment, children will be allocated to two groups by an independent research assistant. Two post-treatment protocols are as follows.

Group A - Children are instructed to rinse their teeth with a cup of water containing about 50 ml immediately after SDF treatment. Afterwards, no post-treatment protocol is given to children.

Group B - Children are instructed not to eat and drink for at least 30 minutes. Clinical examinations after 6-months will be conducted to assess whether the caries is arrested. Information on confounding factors, such as oral hygiene habits and the use of other fluoride agents, will be collected through a parental questionnaire at the baseline and 12-months follow-up. The analysis will determine the significance of differences between the percentage of arrested caries at the various follow-ups.

Significance: This study will help determine the optimal post-op treatment in SDF treatment. The study provides an evidence-based protocol for the use of silver diamine fluoride to arrest tooth decay in primary teeth of young children.

ELIGIBILITY:
Inclusion Criteria:

1. 3-5 year old children attending the first to the third year of kindergarten;
2. free from any systemic conditions and generally healthy;
3. parents sign informed consent;
4. having at least 1 tooth with cavitated dentine carious lesion

Exclusion Criteria:

1. are uncooperative to accept oral examination or treatment;
2. have a significant systematic disease or long-term medications;
3. have abnormal dentition.
4. Teeth having signs or symptoms of irreversible pulpitis and non-vitality will be excluded.

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 254 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Caries status | at 12-month follow-up
  The proportion of the soft (active) carious tooth lesion surfaces that harden (arrested) at 12 months of follow-up will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- The university of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun IG, Duangthip D, Lo ECM, Chu CH. The Caries-Arrest Effectiveness of Silver Diamine Fluoride Treatment with Different Post-Treatment Instructions in Preschool Children: A Study Protocol for a Randomized Controlled Trial. Dent J (Basel). 2023 Jun 5;11(6):145. doi: 10.3390/dj11060145. PMID 37366668